CLINICAL TRIAL: NCT04742894
Title: Neural Bases of Vocal Sensorimotor Impairment in Aphasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Dr. Roozbeh Behroozmand, Associate Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-24-325; R01DC018523 (NIH)
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aphasia Group (Experimental)
  Interventions: Behavioral: Visual Feedback Training
- Control Group (Experimental)
  Interventions: Behavioral: Visual Feedback Training

INTERVENTIONS:
Behavioral: Visual Feedback Training — Participants will be trained to work with a computer setup to control the position of a visual cursor on the screen using their speech while their auditory feedback is altered. The goal of the training is to help improve speech production and motor control ability.

SUMMARY:
Aphasia is the most common type of post-stroke communication disorder characterized by deficits in speech comprehension, production and control. While recovery can be promoted with speech therapy, improvement remains modest and typically requires a large number of sessions contributing to rising health care costs. Traditional aphasia therapy focus on enhancing speech motor output; however, recent evidence suggests that the auditory feedback also plays a critical role in fluent speech. Therefore, a key step toward refining treatment strategies is to develop objective biomarkers that can probe the integrity of sensorimotor mechanisms of speech auditory feedback and identify their impaired function in patients with post-stroke aphasia. This study aims to examine the behavioral, neurophysiological (EEG), and neuroimaging (fMRI) biomarkers of speech impairment following stroke with focus on understanding the role of auditory feedback for speech production and control. We plan to test individuals with post-stroke aphasia and a matched neuroptypical control group during different speech production tasks under the altered auditory feedback paradigm. In addition, we aim to examine the effect of audio-visual feedback training on enhancing communication ability during speech. These biomarkers will be combined with existing lesion-symptom-mapping data in the aphasic group in order to identify the patterns of brain damage and diminished structural connectivity within the auditory-motor areas of the left hemisphere that predict impaired sensorimotor processing of speech in aphasia. The long-term goal of this research is to develop a model for identifying the source of sensorimotor deficit and improve diagnosis and targeted treatment of speech disorders in aphasia.

ELIGIBILITY:
Inclusion Criteria:

* A total of 50 individuals with aphasia due to chronic left hemisphere stroke (> 6 months post-stroke) and 50 age- and gender-matched healthy control subjects will be recruited in this study. The general inclusion criteria for all subjects include: age range 21-75 years, right-handed, and native speaker of English. The aphasic subjects have previously undergone neuro-psychological speech/language testing and have been diagnosed with one type of aphasia (e.g., Broca's, Wernicke's, conduction or anomic). Subjects in the control group will meet the inclusion criteria with having normal voice, speech, language, and hearing function and no history of neurological and psychiatric disorder. We expect that a significant proportion of aphasic patients will show symptoms associated with Apraxia of Speech (AOS) or dysarthria; however, these patients will not be excluded unless their deficits will preclude them from performing the experimental tasks.

Exclusion Criteria:

* Subjects with moderate to severe hearing, memory, and/or cognitive impairments will be excluded for both groups. In addition, subjects with history of peripheral laryngeal disorders (e.g., paresis or vocal fold paralysis) will be excluded. Subjects will undergo safety screening and will be excluded if there are any factors counter-indicative for EEG and/or MRI scanning.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-11 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Speech Production and Motor Control Ability | 2 weeks
  Participants accuracy in using their speech for controlling the visual cursor will be assessed via measuring their deviation from hitting a pre-defined target on the screen.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California Irvine, Irvine, California
  - University of South Carolina, Columbia, South Carolina
  - The University of Texas at Dallas, Richardson, Texas

DOCUMENTS (1):
  • Informed Consent Form (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT04742894/ICF_000.pdf